CLINICAL TRIAL: NCT06112353
Title: Sugammadex VS Neostigmine and Glycopyrrolate Reversal of Neuromuscular Relaxation For Time to Return of Bowel Function After Bowel Resection: Prospective, Randomized, Triple-blinded Clinical Trial For Quality Improvement
Brief Title: Neuromuscular Blockade Comparison for GI-2 Recovery After Bowel Resection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Robert Ryan Field, Associate Clinical Professor, Dept of Anesthesiology & Perioperative Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2295; Field 100931 (Other: Merck Investigator Initiated Studies Program (MISP))
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-05

CONDITIONS: Intestinal Disease
Keywords: Laparoscopic Bowel Resection; Sugammadex; Neostigmine; Glycopyrrolate; GI-2
MeSH Terms: conditions — Intestinal Diseases | interventions — Neostigmine; Glycopyrrolate; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Neostigmine plus Glycopyrrolate (Active Comparator): 0.07 mg/kg Neostigmine plus 0.014 mg/kg glycopyrrolate
  2 syringes numbered 1 and 2
  1. Syringe #1: Glycopyrrolate
  2. Syringe #2: Neostigmine
  Interventions: Drug: Neostigmine Injectable Solution
- Sugammadex (Active Comparator): 2.0 mg/kg of Sugammadex plus saline equivalent
  2 syringes numbered 1 and 2
  1. Syringe #1: 0.9% sodium chloride
  2. Syringe #2: : full Sugammadex dose + 0.9 sodium chloride (QS to match volume)
  Interventions: Drug: Sugammadex injection

INTERVENTIONS:
Drug: Neostigmine Injectable Solution — Examine GI-2 recovery
  Other Names: Neostigmine plus Glycopyrrolate; Group B
  Arms: Neostigmine plus Glycopyrrolate
Drug: Sugammadex injection — Examine GI-2 recovery
  Other Names: Sugammadex; Group A
  Arms: Sugammadex

SUMMARY:
The purpose of this research study is to see the outcome of Sugammadex versus Neostigmine with Glycopyrrolate in colorectal surgery as it relates to its effects on post-surgical time (in hours) to first bowel movement and tolerance for solid food (GI-2 recovery) following bowel resection surgery

DETAILED DESCRIPTION:
Neuromuscular blocking agents are essential during surgical procedures to paralyze the body to avoid unnecessary movement during surgery. There are various medications, such as Sugammadex that are later used to reverse the effects of the neuromuscular blockade. The U.S. performs approximately 320,000 colectomies per year for benign and malignant conditions such as Ulcerative Colitis (UC). Bowel resection surgery removes a portion of small or large intestine. Currently, there is little available prospective outcomes data regarding the use of Sugammadex versus Neostigmine with Glycopyrrolate in colorectal surgery as it relates to its effects on post-surgical time (hour) to first bowel movement and tolerance for solid food (aka GI-2 recovery) following bowel resection surgery. The study team will be conducting a randomized triple-blind study (patient's assigned group is hidden from the patient, provider, and research team). Randomization is created by using an electronic randomizer. Upon consent, the patient's assignment (per the randomizer) will be submitted to the Investigational Drug Service (IDS) Pharmacy by a department employee with no direct patient interaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Laparoscopic bowel resection surgery under general anesthesia with nondepolarizing neuromuscular blockade with rocuronium or vecuronium, and requiring inpatient admission

Exclusion Criteria:

* Allergy to Rocuronium, Vecuronium, or Sugammadex
* Bowel resection surgery requiring an ostomy
* No severe valvulopathy, no systolic heart failure with reduced ejection fraction (HFrEF), no coronary artery disease with positive stress test for ischemic regional wall motion abnormality
* No autoimmune pulmonary disease, no severe pulmonary fibrosis, no severe pulmonary hypertension, no COPD with requirement of home oxygen, no pulmonary cancer of primary or metastatic origin
* Creatinine Clearance (CrCl) of less than 30
* Pregnancy
* Incapable of providing consent or understanding the research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
GI-2 Recovery | Up to 24 hours post surgery
  GI-2 recovery as defined as hour to first bowel movement and toleration of oral diet

SECONDARY OUTCOMES:
Cost of Stay | From hospital admission to discharge, up to 30 days
  Total cost of surgical stay
Length of Stay | From hospital admission to discharge, up to 60 days
  Total time patient is at hospital
Morbidity & Mortality Rate | 30 days post surgery
  Symptomatic disease presence and death
Number of Participants Experiencing Post Reversal Bradycardia | Post surgically but prior to PACU discharge, up to 24 hours
  Slowed heart rate following reversal
Duration of PACU Stay | From surgical end time to PACU discharge, up to 24 hours
  Time in PACU, not owing to bed availability
Time to Out of Bed | Up to 24 hours post surgery
  Time for patient to be able to get out of bed and walk post surgically
Amount of Fluid Administration | Intraoperative
  IV fluid administration during surgery
Presence of Bowel Adhesion | Intraoperative
  Scar tissue found in bowels
Number of Participants Experiencing PONV | Postoperative to discharge, up to 1 week
  Post operative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Field, MD, Principal Investigator — Associate Clinical Professor
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hristovska AM, Duch P, Allingstrup M, Afshari A. Efficacy and safety of sugammadex versus neostigmine in reversing neuromuscular blockade in adults. Cochrane Database Syst Rev. 2017 Aug 14;8(8):CD012763. doi: 10.1002/14651858.CD012763. PMID 28806470
- [Background] Briggs A, Goldberg J. Tips, Tricks, and Technique for Laparoscopic Colectomy. Clin Colon Rectal Surg. 2017 Apr;30(2):130-135. doi: 10.1055/s-0036-1597313. PMID 28381944
- [Background] Deyhim N, Beck A, Balk J, Liebl MG. Impact of Sugammadex Versus Neostigmine/Glycopyrrolate on Perioperative Efficiency. Clinicoecon Outcomes Res. 2020 Jan 31;12:69-79. doi: 10.2147/CEOR.S221308. eCollection 2020. PMID 32099426
- [Background] Gray PJ, Goldwag JL, Eid MA, Sacks OA, Wilson LR, Wilson MZ, Ivatury SJ. Does Bowel Function Change After Colectomy for Colon Malignancy? J Surg Res. 2021 Feb;258:283-288. doi: 10.1016/j.jss.2020.09.003. Epub 2020 Oct 8. PMID 33039637
- [Background] Bhurwal A, Minacapelli CD, Patel A, Mutneja H, Goel A, Shah I, Bansal V, Brahmbhatt B, Das KM. Evaluation of a U.S. National Cohort to Determine Utilization in Colectomy Rates for Ulcerative Colitis Among Ethnicities. Inflamm Bowel Dis. 2022 Jan 5;28(1):54-61. doi: 10.1093/ibd/izab020. PMID 33534892
- [Background] Ludwig K, Enker WE, Delaney CP, Wolff BG, Du W, Fort JG, Cherubini M, Cucinotta J, Techner L. Gastrointestinal tract recovery in patients undergoing bowel resection: results of a randomized trial of alvimopan and placebo with a standardized accelerated postoperative care pathway. Arch Surg. 2008 Nov;143(11):1098-105. doi: 10.1001/archsurg.143.11.1098. PMID 19015469
- [Background] Deljou A, Soleimani J, Sprung J, Schroeder DR, Weingarten TN. Effects of Reversal Technique for Neuromuscular Paralysis on Time to Recovery of Bowel Function after Craniotomy. Am Surg. 2023 May;89(5):1605-1609. doi: 10.1177/00031348211058631. Epub 2022 Jan 5. PMID 34986061
- [Background] Booij LH, van Egmond J, Driessen JJ, de Boer HD. In vivo animal studies with sugammadex. Anaesthesia. 2009 Mar;64 Suppl 1:38-44. doi: 10.1111/j.1365-2044.2008.05869.x. PMID 19222430